CLINICAL TRIAL: NCT02700399
Title: Randomized Crossover Study of Pulse Pressure on Respectively Tilt Table With Integrated Stepping Function (Erigo®) and Traditional Tilt Table in Adult Patients With Acquired Brain Injury
Brief Title: Study of Pulse Pressure During Tilttable and Erigo® in Adult Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SSK01
Record Dates: First submitted 2016-02-05; First posted 2016-03-07 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Brain Injuries; Hypotension, Orthostatic; Syncope
Keywords: Rehabilitation
MeSH Terms: conditions — Brain Injuries; Hypotension, Orthostatic; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erigo® First (Other): Erigo® 0 - 60 degrees - Wash out period (min 30 minutes, max 120 minutes) - Traditional Tilt table 0 - 60 degrees
  Step frequency on Erigo® = 48
  Interventions: Device: Erigo® Hocoma; Device: Traditional tilt table from Rehab-Care
- Traditional first (Other): Traditional Tilt table 0 - 60 degrees - Wash out period (min 30 minutes, max 120 minutes) - Erigo® 0 - 60 degrees
  Step frequency on Erigo® = 48
  Interventions: Device: Erigo® Hocoma; Device: Traditional tilt table from Rehab-Care

INTERVENTIONS:
Device: Erigo® Hocoma — Robotics assisted tilt table, without functional electrical stimulation
Device: Traditional tilt table from Rehab-Care — Traditional tilt table

SUMMARY:
The purpose of this study is to determine if the pulse pressure changes are different whether patients are training in a traditional tilt table as compared to a robotic assisted tilt table, which induces leg movement.

DETAILED DESCRIPTION:
The trial takes place in a non private hospital in Denmark. Patients are recruited from two wards treating patients with severe brain injury, and all patients admitted in the study period are considered in regards to inclusion or exclusion. Patients are included via closest relatives accept, and the patients GP(General Practitioner). Any adverse effect or event will be reported to the local ethics committee. All data will be collected simultaneously with the interventions. Some data will be directly recorded via monitor output, and some data will be directly inputted in Epidata, while trial takes place.

Sample size has been calculated to be between 10 and 60 individuals depending on the actual difference. Beyond 60 included individuals the clinical relevance of a statistical significant result is no longer apparent. If any individual variables are noncomplete, an analysis of the subjects with missing data, will be undertaken.

The statistical analyses planned follows the general crossover design using an approach considering 2 treatment and 2 periods. Patients are cluster randomized in clusters of 4, to be treated with one or the other intervention first.

Intervention A:

Traditional tilt table. measurements at 0 degrees 30 deg. 60. deg. and at return to 0 deg.

Intervention B:

Erigo® tilttable, with measurements as in intervention A. During the intervention the step frequency of the Erigo® i set at 48 steps/min.

Between the two periods a wash out period of at least ½ hour and maximum 2 hours are planned.

Primary outcome is derived from noninvasive BP measurements.

ELIGIBILITY:
Inclusion Criteria:

* Already being treated with traditional tilttable and must be able to benefit from Erigo® treatment from a clinicians view
* Acquired brain injury as primary diagnose
* Must have Rancho Los Amigo Scale score of minimum 1 to maximum 6 on the day of inclusion

Exclusion Criteria:

* Not on mechanical ventilation
* New cerebral, cardiological or other medical problems/emergencies between the 2 interventions
* Change in cardiac medications between interventions
* Patient must not have independent gait function immediately before trial
* must not have EFA(Early Functional abilities) part score > 4 in the section "Standing", assessed by the treating physiotherapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Non Invasive Blood Pressure(NIBP) | Measured at: Baseline in supine on tilttable, 60 seconds after 30 degrees rise of tilttable, 60 seconds after 60 degrees tilt is reached. Again 60 seconds after return to 0 degrees tilt with patient still in supine position on tilttable..

SECONDARY OUTCOMES:
Patient reported comfort: The difference in prevalence of both acceptable- and not acceptable patient comfort between the Erigo and the conventional tilt-table. | Question is asked within 5 minutes after 60 degrees NIBP measurement
  Due to the included patients level of consciousness, comfort is reported as the treating therapists subjective evaluation of patients answers to standardized visual and audial question.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Prof.MD DMSc, Study Director — Regionshospitalet Hammel Neurocenter
Locations (1):
- Regionshospitalet Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No